CLINICAL TRIAL: NCT03001297
Title: A Phase 1 Randomized, Blinded, Placebo-controlled Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Single-Ascending Doses of MEDI5884 in Healthy Volunteers
Brief Title: Phase 1, Single Dose Study to Evaluate Safety, Pharmacokinetics, and Pharmacodynamics of MEDI5884
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D7870C00001
Record Dates: First submitted 2016-11-23; First posted 2016-12-23 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Healthy Volunteers
Keywords: atherosclerosis; acute coronary syndrome; MEDI5884
MeSH Terms: conditions — Atherosclerosis; Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- MEDI5884 Dose 1 (Experimental): Participants will receive single dose of MEDI5884 Dose 1 injection SC on Day 1.
  Interventions: Biological: MEDI5884 Dose 1
- Placebo (Placebo Comparator): Placebo will be administered subcutaneously (SC).
  Interventions: Biological: Placebo
- MEDI5884 Dose 2 (Experimental): Participants will receive single dose of MEDI5884 Dose 2 injection SC on Day 1.
  Interventions: Biological: MEDI5884 Dose 2
- MEDI5884 Dose 3 (Experimental): Participants will receive single dose of MEDI5884 Dose 3 injection SC on Day 1.
  Interventions: Biological: MEDI5884 Dose 3
- MEDI5884 Dose 4 (Experimental): Participants will receive single dose of MEDI5884 Dose 4 injection SC on Day 1.
  Interventions: Biological: MEDI5884 Dose 4

INTERVENTIONS:
Biological: Placebo — Participants will receive single dose of placebo matched MEDI5884 injection SC on Day 1
  Arms: Placebo
Biological: MEDI5884 Dose 1 — Participants will receive single dose MEDI5884 Dose 1 injection SC on Day 1.
  Arms: MEDI5884 Dose 1
Biological: MEDI5884 Dose 2 — Participants will receive single dose MEDI5884 Dose 2 injection SC on Day 1
  Arms: MEDI5884 Dose 2
Biological: MEDI5884 Dose 3 — Participants will receive single dose MEDI5884 Dose 3 injection SC on Day 1
  Arms: MEDI5884 Dose 3
Biological: MEDI5884 Dose 4 — Participants will receive single dose MEDI5884 Dose 4 injection SC on Day 1
  Arms: MEDI5884 Dose 4

SUMMARY:
A Phase 1, single dose study with 4 cohorts of ascending doses and an optional Japanese cohort designed to evaluate the safety, pharmacokinetics, and pharmacodynamics of MEDI5884 in healthy volunteers

DETAILED DESCRIPTION:
This is a first time in human, phase 1, randomized, blinded, placebo-controlled study to evaluate the safety, pharmacokinetics and pharmacodynamics of single ascending subcutaneous doses of MEDI5884 in healthy volunteers (age 18-55). The study consists of 4 cohorts of increasing doses (8 subjects each) and an optional Japanese American cohort (24 subjects) for a total of 56 healthy subjects. The decision whether or not to dose escalate will be based upon data review by the Dose Escalation Committee. Subjects will be randomized 3:1 to MEDI5884 or placebo. Following screening, the study consists of a 3 day inpatient stay and follow up visits. The number of follow up visits depend on the cohort assigned.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged 18-55 years
* Must provide written informed consent
* Ability and willingness to adhere to the protocol
* BMI 18-30kg/m2
* Females not of childbearing potential
* Males must practice 2 effective contraceptive measures if sexually active
* Japanese descent for the Japanese cohort

Exclusion Criteria:

* Any concurrent condition that in the opinion of the investigator would interfere with the evaluation of the investigational product
* History or presence of gastrointestinal, renal, or hepatic disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs
* Abnormal lab values, physical exam, vital signs
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks prior to dosing
* Positive Hepatitis B, Hepatitis C or HIV test
* Receipt of investigational therapy with 4 months from screening
* Current or previous use of systemic corticosteroids 60 days prior to dosing or lipid lowering medications 28 days prior to dosing
* Abnormal ECG
* Recent plasma or blood donation
* Positive drug or alcohol screen.
* Current smoker

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events as a measure of safety and tolerability of MEDI5884 | Baseline until last follow-up visit, assessed up to 90 days post dose depending on cohort.
  Treatment emergent adverse events (TEAEs) and serious adverse events (TESAEs)
Number of subjects with adverse events as a measure of safety and tolerability of MEDI5884 | Baseline until last follow-up visit, assessed up to 90 days post dose depending on cohort.
  12 lead electrocardiogram (ECG) including RR (The time between corresponding points on 2 consecutive R waves on ECG), PR (ECG interval measured from the onset of the P wave to the onset of the QRS complex) , QRS (ECG interval measured from the onset of the QRS complex to the J point) , QT (ECG interval measured from the onset of the QRS complex to the end of the T wave), and QTc (QT interval corrected for heart rate) intervals
Number of subjects with adverse events as a measure of safety and tolerability of MEDI5884 | Baseline until last follow-up visit, assessed up to 90 days post dose depending on cohort.
  Vital signs (systolic and diastolic blood pressure, pulse rate, temperature, and respiratory rates)
Number of subjects with adverse events as a measure of safety and tolerability of MEDI5884 | Baseline until last follow-up visit, assessed up to 90 days post dose depending on cohort.
  Clinical laboratory assessments (serum chemistry, hematology, and urinalysis)
HDL-Cholesterol over time | Baseline until last follow-up visit, assessed up to 90 days post dose depending on cohort.
  HDL-Cholesterol over time

SECONDARY OUTCOMES:
Lipoprotein particle size | Cohort 1: 28 days post dosing, Cohort 2: 45 days post dosing , Cohort 3: 60 days post dosing, Cohort 4: 90 days posting dosing, Optional Japanese American cohort: 60 days posting dosing
  Lipoprotein particle size
Lipoprotein particle number | Cohort 1: 28 days post dosing, Cohort 2: 45 days post dosing , Cohort 3: 60 days post dosing, Cohort 4: 90 days posting dosing, Optional Japanese American cohort: 60 days posting dosing
  Lipoprotein particle number
Levels of total cholesterol | Cohort 1: 28 days post dosing, Cohort 2: 45 days post dosing , Cohort 3: 60 days post dosing, Cohort 4: 90 days posting dosing, Optional Japanese American cohort: 60 days posting dosing
  Levels of total cholesterol
Non-HDL-Cholesterol | Cohort 1: 28 days post dosing, Cohort 2: 45 days post dosing , Cohort 3: 60 days post dosing, Cohort 4: 90 days posting dosing, Optional Japanese American cohort: 60 days posting dosing
  Non-HDL-Cholesterol
Low-density lipoprotein cholesterol (direct and Friedewald equation) | Cohort 1: 28 days post dosing, Cohort 2: 45 days post dosing , Cohort 3: 60 days post dosing, Cohort 4: 90 days posting dosing, Optional Japanese American cohort: 60 days posting dosing
  Low-density lipoprotein cholesterol (direct and Friedewald equation)
Very low-density lipoprotein cholesterol | Cohort 1: 28 days post dosing, Cohort 2: 45 days post dosing , Cohort 3: 60 days post dosing, Cohort 4: 90 days posting dosing, Optional Japanese American cohort: 60 days posting dosing
  Very low-density lipoprotein cholesterol
Triglycerides | Cohort 1: 28 days post dosing, Cohort 2: 45 days post dosing , Cohort 3: 60 days post dosing, Cohort 4: 90 days posting dosing, Optional Japanese American cohort: 60 days posting dosing
  Triglycerides
Apolipoprotein B | Cohort 1: 28 days post dosing, Cohort 2: 45 days post dosing , Cohort 3: 60 days post dosing, Cohort 4: 90 days posting dosing, Optional Japanese American cohort: 60 days posting dosing
  Apolipoprotein B
Apolipoprotein A1 | Cohort 1: 28 days post dosing, Cohort 2: 45 days post dosing , Cohort 3: 60 days post dosing, Cohort 4: 90 days posting dosing, Optional Japanese American cohort: 60 days posting dosing
  Apolipoprotein A1
MEDI5884 serum concentration: maximum observed concentration | Post dose on Days 1, 2, 3, 7, 14, 21, 28, 45 (cohorts 2-4 and Japanese American), 60 (cohorts 3, 4 and Japanese American), 75 (cohort 4), and 90 (cohort 4)
  MEDI5884 serum concentration: maximum observed concentration
MEDI5884 serum concentration: time to maximum observed concentration | Post dose on Days 1, 2, 3, 7, 14, 21, 28, 45 (cohorts 2-4 and Japanese American), 60 (cohorts 3, 4 and Japanese American), 75 (cohort 4), and 90 (cohort 4)
  MEDI5884 serum concentration:
  time to maximum observed concentration
MEDI5884 serum concentration: area under the concentration time curve | Post dose on Days 1, 2, 3, 7, 14, 21, 28, 45 (cohorts 2-4 and Japanese American), 60 (cohorts 3, 4 and Japanese American), 75 (cohort 4), and 90 (cohort 4)
  MEDI5884 serum concentration: area under the concentration time curve
MEDI5884 serum concentration: terminal half-life | Post dose on Days 1, 2, 3, 7, 14, 21, 28, 45 (cohorts 2-4 and Japanese American), 60 (cohorts 3, 4 and Japanese American), 75 (cohort 4), and 90 (cohort 4)
  MEDI5884 serum concentration:
  terminal half-life
Anti-drug antibody | Cohort 1: 28 days post dosing, Cohort 2: 45 days post dosing , Cohort 3: 60 days post dosing, Cohort 4: 90 days posting dosing, Optional Japanese American cohort: 60 days posting dosing
  Anti-drug antibody

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Glendale, California, United States